CLINICAL TRIAL: NCT02276222
Title: A Randomized, Open-Label, Active-Controlled, Parallel-Group, Multicenter, Long-Term Safety Trial of Treatment With Nebulized SUN-101 in Patients With COPD: GOLDEN-5 (Glycopyrrolate for Obstructive Lung Disease Via Electronic Nebulizer)
Brief Title: A Long-Term Safety Trial of Treatment With Nebulized SUN-101 in Patients With COPD
Acronym: GOLDEN-5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunovion Respiratory Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUN101-303
Record Dates: First submitted 2014-10-14; First posted 2014-10-28 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Nebulizers and Vaporizers; Glycopyrrolate; Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SUN-101 50 mcg BID eFlow (CS) nebulizer (Experimental): SUN-101 (Glycopyrrolate) 50 mcg twice daily (BID) via eFlow Closed System (CS) nebulizer
  Interventions: Drug: SUN-101 50 mcg BID eFlow (CS) nebulizer
- Spiriva 18 mcg QD Handihaler (Active Comparator): Spiriva (tiotropium) 18 mcg once daily (QD) via Handihaler
  Interventions: Drug: Spiriva® 18 mcg QD Handihaler

INTERVENTIONS:
Drug: SUN-101 50 mcg BID eFlow (CS) nebulizer — SUN-101 (Glycopyrrolate) 50 mcg twice daily (BID) via eFlow Closed System (CS) nebulizer
  Other Names: Glycopyrrolate
  Arms: SUN-101 50 mcg BID eFlow (CS) nebulizer
Drug: Spiriva® 18 mcg QD Handihaler — Spiriva (tiotropium) 18 mcg once daily (QD) via Handihaler
  Other Names: (tiotropium)
  Arms: Spiriva 18 mcg QD Handihaler

SUMMARY:
This is a long-term safety trial of 48 weeks. Eligible subjects will enter the 48-week, open-label treatment period to receive one of two treatments (SUN-101 given as 50 mcg twice a day or Spiriva® [tiotropium] given as 18 mcg once a day).

DETAILED DESCRIPTION:
This is a Phase 3, randomized, open-label, active-controlled, parallel-group, multicenter, long-term safety trial of 48 weeks of treatment with nebulized SUN-101 using an Investigational eFlow® Closed System (CS) nebulizer or Spiriva in approximately 1050 subjects with chronic obstructive pulmonary disease (COPD) according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD 2014) guidelines.

Eligible subjects will enter the 48-week, open-label treatment period following randomization to receive one of two treatments (SUN-101 given as 50 mcg BID or Spiriva® [tiotropium] given as 18 mcg QD).

The hypothesis for this study is that the incidence of treatment-emergent adverse events reported over the course of 48 weeks of treatment by subjects randomized to SUN-101 is numerically similar to the incidence of treatment-emergent adverse events reported over the course of 48 weeks of treatment by subject randomized to Spiriva (tiotropium).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age ≥ 40 years, inclusive.
2. A clinical diagnosis of COPD according to the GOLD 2014 guidelines.
3. Current smokers or ex-smokers with at least 10 pack-year smoking history (eg, at least 1 pack/day for 10 years, or equivalent).
4. Post-bronchodilator (following inhalation of ipratropium bromide) FEV1 < 80% of predicted normal and > 0.7 L during Screening (Visit 1).
5. Post-bronchodilator (following inhalation of ipratropium bromide) FEV1/FVC ratio < 0.70 during Screening (Visit 1).
6. Ability to perform reproducible spirometry according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) guidelines (2005).
7. Subject, if female ≤ 65 years of age and of child bearing potential, must have a negative serum pregnancy test at Visit 1. Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study and must use an acceptable method of birth control: a) an oral contraceptive, an intrauterine device (IUD), implantable contraceptive, transdermal or injectable contraceptive for at least 1 month prior to entering the study with continued use throughout the study and for thirty days following participation; b) barrier method of contraception, e.g., condom and /or diaphragm with spermicide while participating in the study; and/or c) abstinence..
8. Willing and able to provide written informed consent.
9. Willing and able to attend all study visits and adhere to all study assessments and procedures.

Exclusion Criteria:

1. Severe comorbidities including unstable cardiac or pulmonary disease or any other medical conditions that would, in the opinion of the Investigator, preclude the subject from safely completing the required tests or the study, or is likely to result in disease progression that would require withdrawal of the subject.
2. Concomitant clinically significant respiratory disease other than COPD (eg, asthma, tuberculosis, bronchiectasis or other non-specific pulmonary disease).
3. Recent history of COPD exacerbation requiring hospitalization or need for increased treatments for COPD within 6 weeks prior to Screening (Visit 1).
4. Use of daily oxygen therapy > 12 hours per day.
5. Respiratory tract infection within 6 weeks prior to Screening (Visit 1).
6. Use of systemic steroids within 3 months prior to Screening (Visit 1).
7. History of malignancy of any organ system, treated or untreated within the past 5 years, with the exception of localized basal cell carcinoma of the skin.
8. Prolonged QTc (> 450 msec for males and > 470 msec for females) during Screening (Visit 1), or history of long QT syndrome.
9. History of or clinically significant ongoing bladder outflow obstruction or history of catheterization for relief of bladder outflow obstruction within the previous 6 months.
10. History of narrow angle glaucoma.
11. History of hypersensitivity or intolerance to aerosol medications.
12. Recent documented history (within the previous 3 months) of substance abuse.
13. Significant psychiatric disease that would likely result in the subject not being able to complete the study, in the opinion of the Investigator.
14. Participation in another investigational drug study where drug was received within 30 days prior to Screening (Visit 1) or current participation in another investigational drug trial, including a SUN-101 study.
15. Previously received SUN-101 (active treatment; formerly known as EP-101).
16. Contraindicated for treatment with, or having a history of reactions/ hypersensitivity to anticholinergic agents, beta2 agonists, or sympathomimetic amines.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1087 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Respiratory Medical Director, Study Director — Sunovion Respiratory Development
Locations (118):
- United States (83):
  - SEC Lung LLC, Andalusia, Alabama
  - Achieve Clinical Research LLC, Birmingham, Alabama
  - Jasper Summit Research LLC, Jasper, Alabama
  - Clinical Research Advantage, Inc.lEast Valley Family Physicians, PLC, Chandler, Arizona
  - Desert Sun Clinical Research LLC, Tucson, Arizona
  - Allianz Research Institute, Inc., Fountain Valley, California
  - Research Center of Fresno, Inc., Fresno, California
  - California Research Medical Group, lnc., Fullerton, California
  - Southern California Institute For Respiratory Diseases, Inc., Los Angeles, California
  - Integrated Research Group, Inc, Riverside, California
  - Institute of Healthcare Assessments Inc., San Diego, California
  - Waterbury Pulmonary Associates, LLC, Waterbury, Connecticut
  - Tampa Bay Clinical Research Center, Brandon, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - Avail Clinical Research, llC, DeLand, Florida
  - The Community Research of South Florida, Hialeah, Florida
  - AppleMed Research, Inc, Miami, Florida
  - Research Institute of South Florida, Inc, Miami, Florida
  - Clinical Trials of Florida, LLC, Miami, Florida
  - Florida Institute For Clinical Research, LLC, Orlando, Florida
  - Ribo Research, LLC dba Peninsula Research, Inc., Ormond Beach, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Vero Lung Center, Vero Beach, Florida
  - Gwinnett Biomedical Research, Lawrenceville, Georgia
  - H.C. Research LLC, Coeur d'Alene, Idaho
  - Evanston Premier Healthcare Research LLC, Evanston, Illinois
  - Asthma and Allergy Center of Chicago SC, River Forest, Illinois
  - LaPorte County Institute For Clinical Research, Michigan City, Indiana
  - Buynak Clinical Research, P.C., Valparaiso, Indiana
  - Abraham Research, PLLC, Fort Mitchell, Kentucky
  - Kentucky Lung Clinics, PSC, Hazard, Kentucky
  - Bendel Medical Research Center, LLC, Lafayette, Louisiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Howard County Center for Lung and Sleep Medicine, LLC, Columbia, Maryland
  - Pulmonary and Critical Care Associates of Baltimore, Towson, Maryland
  - Cadillac Clinical Research LLC, Cadillac, Michigan
  - Pulmonary Research Institute of Southeast Michigan, Livonia, Michigan
  - Minnesota Lung Center, Edina, Minnesota
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Minnesota Lung Center, Minneapolis, Minnesota
  - Minnesota Lung Center, Woodbury, Minnesota
  - Midwest Chest Consultants PC, Saint Charles, Missouri
  - CARE Clinical Research, St Louis, Missouri
  - Midwest Clinical Research LLC, St Louis, Missouri
  - The Clinical Research Center, St Louis, Missouri
  - Somnos Laboratories, Inc d/b/a Somnos Clinical Research, Lincoln, Nebraska
  - Clinical Research Advantage Inc, Las Vegas, Nevada
  - Delaware Valley Clinical Research, LLC, Marlton, New Jersey
  - Atlantic Research Center, LLC, Ocean City, New Jersey
  - Pulmonary and Allergy Associates, PA, Summit, New Jersey
  - ISA Clinical Research, Jamaica, New York
  - American Health Research, Inc., Charlotte, North Carolina
  - ARSM Research, Huntersville, North Carolina
  - Clinical Research of Lake Norman, Huntersville, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - IVA Researcb, Cincinnati, Ohio
  - Remington Davis Inc, Columbus, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Sunstone Medical Research, L.LC, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Lowcountry Lung and Critical Care, PA, Charleston, South Carolina
  - Easley Clinical Research, Easley, South Carolina
  - Palmetto Medical Research Associates, Easley, South Carolina
  - Gaffney Pharmaceutical Research, Gaffney, South Carolina
  - Spectrum Medical Research, LLC, Gaffney, South Carolina
  - Greenville Pharmaceutical Research, Inc., Greenville, South Carolina
  - Upstate Pharmaceutical Research, Inc., Greenville, South Carolina
  - DeGarmo Institute of Medical Research, Greer, South Carolina
  - Clinical Research of Charleston, Mt. Pleasant, South Carolina
  - Hope Clinical Research, Seneca, South Carolina
  - S. Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - CU Pharmaceutical Research, Union, South Carolina
  - New Phase Clinical Research & Development, Knoxville, Tennessee
  - Corsicana Medical Research, PLLC, Corsicana, Texas
  - Pioneer Research Solutions, Inc, Houston, Texas
  - Alamo Clinical Research Associates, San Antonio, Texas
  - Pulmonary Consultants PLLC, Tacoma, Washington
- Czechia (9):
  - Medicentrum Beroun s.r o., Beroun
  - MediTrial, s.r.o Internf a pneumoloqicka ambulance, Jindřichův Hradec
  - Nemocnice Kyjov, p.o., Kyjov
  - Plicni ambulance, Neratovice
  - MephaCentrum, a s Plicni oddeleni, Ostrava - Poruba
  - MephaCentrum, a.s., Ostrava-Poruba
  - PNEUMa-HOST s LO., Prague
  - PLiCNI AMBULANCE ROKYCANY, s.r o., Rokycany
  - Hrudnf ambulance s.r.o., Žatec
- Hungary (12):
  - Dr. Kenessey Albert Korhaz-Rendetointezet, TOd6gy6gyaszati, Balassagyarmat
  - Csornai Margit Korhaz, TOd6gy6gyaszat, Csorna
  - Kenezy Gyula Korhaz es Rendelomtezet, Klinikai Farmakologiai, Debrecen
  - Veszprern Megyei Tudbgyogyintezet, Farkasgyepű
  - Somogy Megyei Kaposi M6r Oktat6 Korhaz, Tudoqondozo, Kaposvár
  - Lumniczer Sandor Korhaz as Rendelointezet, Tudoqondozo, Kapuvár
  - Selye Janos Korhaz es Rendelointezet, Tud6gy6gyaszati Szakrendeles, Komárom
  - Szakorvosi Rendelointezet Monor, Tudoqondozo, Monor
  - Revamed Eqeszsequqyi Szolqaltato Kft., Nyíregyháza
  - Si6fok Kornaz-Rendelointezet, Tudoqondozo, Siófok
  - Farmakontroll Egeszsegugyi Szolqaltato Bt, Százhalombatta
  - Csonqrad Megyei Mellkasi Beteqseqek Szakkorhaza, Tudoqondozo lntezet, Szeged
- Russia (14):
  - Territorial SBI of Healthcare <Territorial Clinical Hospital>, Barnaul
  - FSBI Far Eastern Research Centre ofPhysiology and Pathology of Breathing of Siberian branch of RAMS, Blagoveshchensk
  - SBI of Healthcare Regional Clinical Hospital #4 City consultative department for pulmonological patientsr, Chelyabinsk
  - Municipal Budget Institution of Healthcare (City Clinical Hospital #3 n.a. M.A. Podgorbunsky), Kemerovo
  - FSSI Scientific Research Institute of Complex Cardiovascular Pathology, Kemerovo
  - FSBI, Moscow
  - Non-State Private Institution of Healthcare <Scientific Clinical Center>, Moscow
  - SBI of Healthcare of Nizhny-Novgorod region, Nizhny Novgorod
  - SB1 of Healthcare of Novosibirsk region <Novosibirsk State Regional Clinical Hospital>l, Novosibirsk
  - SBI of Healthcare of Novosibirsk region <Novosibirsk State Regional Clinical Hospital>, Novosibirsk
  - Alliance Biomedical, Russian Group LLC, Saint Petersburg
  - SBEI of HPE <North-West State Medical University n.a. LL Mechnikov>, Saint Petersburg
  - SBr of Helathcareof Yaraslavl region Clinical Hospital of Emervency care n.a.N.V. Solovyev, Yaroslavl
  - Municipal Autonomous Institution (City ClinicalHospital #14), Yekaterinburg

REFERENCES:
- [Result] Ferguson GT, Goodin T, Tosiello R, Wheeler A, Kerwin E. Long-term safety of glycopyrrolate/eFlow(R) CS in moderate-to-very-severe COPD: Results from the Glycopyrrolate for Obstructive Lung Disease via Electronic Nebulizer (GOLDEN) 5 randomized study. Respir Med. 2017 Nov;132:251-260. doi: 10.1016/j.rmed.2017.08.020. Epub 2017 Aug 24. PMID 28919143
- [Derived] Ferguson GT, Kerwin EM, Donohue JF, Ganapathy V, Tosiello RL, Bollu VK, Rajagopalan K. Health-Related Quality of Life Improvements in Moderate to Very Severe Chronic Obstructive Pulmonary Disease Patients on Nebulized Glycopyrrolate: Evidence from the GOLDEN Studies. Chronic Obstr Pulm Dis. 2018 Jun 6;5(3):193-207. doi: 10.15326/jcopdf.5.3.2017.0178. PMID 30584583

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | Spiriva 18 mcg QD Handihaler
Started | 621 | 466
Completed | 436 (one subject withdrew at randomization due to a pre-treatment event prior to being dosed) | 402
Not Completed | 185 | 64
Not completed — Adverse Event | 62 | 11
Not completed — Death | 3 | 4
Not completed — Lack of Efficacy | 13 | 3
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 79 | 33
Not completed — non compliance with study medication | 6 | 2
Not completed — sponsor decision | 0 | 3
Not completed — Lost to Follow-up | 15 | 5
Not completed — Physician Decision | 2 | 1
Not completed — sheduling conflict | 1 | 0
Not completed — subject withdrew after randomization | 1 | 0

BASELINE CHARACTERISTICS:
Population: As noted in the participant flow section, one subject withdrew at randomization due to a pre-treatment event prior to being dosed bringing the population total to 1086 from 1087.
Groups:
- Total: Total of all reporting groups
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | Spiriva 18 mcg QD Handihaler | Total
Number analyzed (Participants) | 620 | 466 | 1086
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 330 | 256 | 586
  >=65 years | 290 | 210 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (8.46) | 63.3 (8.97) | 63.3 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 270 | 206 | 476
  Male | 350 | 260 | 610
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 611 | 457 | 1068
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 27 | 62
  White | 582 | 436 | 1018
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 25 | 21 | 46
  Czechia | 5 | 4 | 9
  Hungary | 34 | 20 | 54
  United States | 556 | 421 | 977
cardiovascular risk (low/high) and categories for high cardiovascular risk [Count of Participants; unit: Participants]
  low cardiovascular risk | 219 | 169 | 388
  high cardiovascular risk | 401 | 297 | 698
  ischemic heart disease | 61 | 44 | 105
  cerebrovascular disease | 28 | 18 | 46
  periheral arterial disease | 39 | 24 | 63
  clinically significant arrhythmia | 22 | 14 | 36
  heart failure | 23 | 9 | 32
  hyertension | 362 | 275 | 637
background long-acting beta (2) agonist (LABA) use [Count of Participants; unit: Participants]
  background LABA use -yes | 267 | 192 | 459
  background LABA use -no | 353 | 274 | 627
Forced expiratory volume in one second (FEV1) [Mean (Standard Deviation); unit: liters] | 1.3399 (0.49604) | 1.3257 (0.50186) | 1.3365 (0.51414)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAE)
Description: A TEAE is any adverse event (AE) that occurred on or after the first dose of study medication, any AE with a missing start date and a stop date on or after the first dose of study medication, or any AE with both a missing start and stop date.
Time Frame: Up to Week 48
Population: Safety population was defined as all subjects who were randomized to treatment and received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | Spiriva 18 mcg QD Handihaler
Number analyzed (Participants) | 620 | 466
participants | 430 | 312

2. Primary Outcome: Percentage of Subjects With Treatment-emergent Adverse Events
Description: as for outcome 1
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | Spiriva 18 mcg QD Handihaler
Number analyzed (Participants) | 620 | 466
percentage of participants | 69.4 | 67.0

3. Primary Outcome: Number of Subjects With Treatment-emergent Serious Adverse Events (SAE)
Description: A treatment emergent serious adverse event (SAE) is any SAE that occurred on or after the first dose of study medication, any SAE with a missing start date and a stop date on or after the first dose of study medication, or any SAE with both a missing start and stop date.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | Spiriva 18 mcg QD Handihaler
Number analyzed (Participants) | 620 | 466
participants | 76 | 49

4. Primary Outcome: Percentage of Subjects With Treatment-emergent Serious Adverse
Description: as for outcome 3
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | Spiriva 18 mcg QD Handihaler
Number analyzed (Participants) | 620 | 466
percentage of participants | 12.3 | 10.5

5. Primary Outcome: Number of Subjects Who Discontinue the Study Due to TEAE
Description: as for outcome 1
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | Spiriva 18 mcg QD Handihaler
Number analyzed (Participants) | 620 | 466
participants | 62 | 13

6. Primary Outcome: Percentage of Subjects Who Discontinue the Study Due to TEAE
Description: as for outcome 1
Time Frame: Up to 48 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | Spiriva 18 mcg QD Handihaler
Number analyzed (Participants) | 620 | 466
percentage of participants | 10.0 | 2.8

7. Secondary Outcome: Number of Subjects With Major Adverse Cardiac Events (MACE), Including Cardiovascular Death, Ischemia/Infarction, and Stroke
Description: All deaths and any other findings suggestive of a potential MACE (including clinically relevant information and SAEs, and all PTs form the SMQs "myocardial infarction", "other ischemic heart disease", "central nervous system hemorrhages and cerebrovascular conditions") were sent to an adjudication committee for review and categorized as CV death, nonfatal MI, and nonfatal stroke. The MACE score was defined as the total number of subjects with CV deaths, nonfatal MIs, and nonfatal strokes. These events were collected from the first date of study medication until the date of last contact.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | Spiriva 18 mcg QD Handihaler
Number analyzed (Participants) | 620 | 466
participants
  MACE score | 3 | 8
  cardiovascular death | 1 | 2
  non-fatal myocardial infarction | 2 | 5
  non-fatal stroke | 0 | 1

8. Secondary Outcome: Percentage of Subjects With Major Adverse Cardiac Events (MACE), Including Cardiovascular Death, Ischemia/Infarction, and Stroke
Description: as for outcome 7
Time Frame: Up to 48 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | Spiriva 18 mcg QD Handihaler
Number analyzed (Participants) | 620 | 466
percentage of participants
  MACE score | 0.5 | 1.7
  cardiovascular death | 0.2 | 0.4
  non-fatal myocardial infarction | 0.3 | 1.1
  non-fatal stroke | 0 | 0.2

9. Secondary Outcome: Incidence Rate Per 1000 Person Years of Subjects With Major Adverse Cardiac Events (MACE), Including Cardiovascular Death, Ischemia/Infarction, and Stroke
Description: as for outcome 7
Time Frame: up to week 48
Population: Incidence rate: TT= Total Time in years. Total Time (TT) is defined as the time from the first date of study drug until the latter of the date of last contact or 30 days after the date of last dose. Incidence Rate (per 1000 person-years) = n/TT x 1000.
Measure: Number; unit: event per 1000 person years
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | Spiriva 18 mcg QD Handihaler
Number analyzed (Participants) | 620 | 466
event per 1000 person years
  MACE score | 6.4 | 20.3
  cardiovascular death | 2.1 | 5.1
  non-fatal myocardial infarction | 4.3 | 12.7
  non-fatal stroke | 0 | 2.5

10. Secondary Outcome: Mean Change From Baseline Over 48 Weeks in Trough FEV1 for All Subjects
Description: Spirometry was performed according to internationally accepted standards. Trough FEV1 was defined as the average of the FEV1 values collected at the end of the dosing interval at each clinic visit. The mean change from baseline in trough FEV1 over the 48 week treatment period is calculated by averaging the trough FEV1 changes from baseline across all study visits while subjects are taking randomized treatment.
  Values affected by other medication use were to be set to missing.
Time Frame: Up to Week 48
Population: Intent to Treat (ITT) Population: all subjects who were randomized to treatment and received at least one dose of study medication. Subjects were analyzed based on the treatment they were randomized to.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | Spiriva 18 mcg QD Handihaler
Number analyzed (Participants) | 620 | 466
liters | 0.1016 (0.00698) | 0.0931 (0.00779)
Statistical Analysis 1: Comparison: SUN-101 50 mcg BID eFlow (CS) Nebulizer vs Spiriva 18 mcg QD Handihaler; Test type: Superiority; p = 0.4041, ANCOVA; Least Squares Mean (SE) = 0.0084, 95% CI 2-sided [-0.0114 to 0.0283], Standard Error of Mean 0.01012

ADVERSE EVENTS:
Time Frame: up to week 48
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | Spiriva 18 mcg QD Handihaler
All-Cause Mortality (participants affected / at risk) | 3/620 | 4/466
Serious Adverse Events (participants affected / at risk) | 76/620 | 49/466
Other Adverse Events (participants affected / at risk) | 195/620 | 133/466
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SUN-101 50 mcg BID eFlow (CS) Nebulizer (N=620) | Spiriva 18 mcg QD Handihaler (N=466)
acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
arterial flutter (Cardiac disorders) | 1 (1) | 0 (0)
cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (2)
cardio respiratory arrest (Cardiac disorders) | 3 (3) | 1 (1)
coronary artery disease (Cardiac disorders) | 3 (3) | 0 (0)
myocardial infraction (Cardiac disorders) | 1 (1) | 1 (1)
verntricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
diplopia (Eye disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
duodenal ulcer, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
chest pain (General disorders) | 1 (1) | 0 (0)
generalized oedema (General disorders) | 1 (1) | 0 (0)
non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
pain (General disorders) | 1 (1) | 0 (0)
pyrexia (General disorders) | 0 (0) | 1 (1)
cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
choleithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
appendicitis (Infections and infestations) | 1 (1) | 1 (1)
bronchitis (Infections and infestations) | 2 (2) | 1 (1)
gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
gastronenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
pheumonia (Infections and infestations) | 8 (8) | 3 (3)
sepsis (Infections and infestations) | 0 (0) | 3 (3)
septic shock (Infections and infestations) | 0 (0) | 1 (1)
systemic candida (Infections and infestations) | 1 (1) | 0 (0)
urinary tract infection (Infections and infestations) | 2 (2) | 1 (3)
urosepsis (Infections and infestations) | 1 (1) | 0 (0)
accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
impacted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
joint effsion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
carcinoid tumor of the apendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
non-hodgkins lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
pancreatic crcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
hashimoto's encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
multile sclerosis relapse (Nervous system disorders) | 0 (0) | 1 (1)
serotonin syndrome (Nervous system disorders) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 1 (1) | 0 (0)
transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
suicidal ideation (Nervous system disorders) | 2 (2) | 0 (0)
renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 14 (15)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
aortic aneurysm (Vascular disorders) | 2 (2) | 1 (2)
arterios clerosis (Vascular disorders) | 0 (0) | 1 (1)
hypertension (Vascular disorders) | 1 (1) | 0 (0)
pluritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SUN-101 50 mcg BID eFlow (CS) Nebulizer (N=620) | Spiriva 18 mcg QD Handihaler (N=466)
nasopharyngitis (Infections and infestations) | 25 (31) | 28 (32)
upper respiratory tract infection (Infections and infestations) | 38 (42) | 25 (28)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 91 (119) | 82 (107)
cough (Respiratory, thoracic and mediastinal disorders) | 73 (78) | 26 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study , the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.